CLINICAL TRIAL: NCT06360471
Title: Fertility Preservation and Pregnancy and Offspring Health Outcomes in Female Cancer Patients: A Multicenter, Prospective, Cohort Study
Brief Title: Fertility Preservation and Pregnancy and Offspring Health Outcomes in Female Cancer
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: FS-FMC
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Fertility Issues; Cancer
Keywords: fertility preservation; cancer
MeSH Terms: conditions — Infertility; Neoplasms | interventions — Fertility Preservation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — the patient blood samples were collected for further study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fertility preservation: patients who choose fertility preservation
  Interventions: Other: fertility preservation
- Observation: patients who choose observation

INTERVENTIONS:
Other: fertility preservation — If a patient have a desire to fertility preservation, oocyte freezing or embryo freezing will be offered.
  Groups: Fertility preservation

SUMMARY:
To explore whether there is a significant difference in the cumulative live birth rate and maternal and child health outcomes between cancer patients who undergo or do not undergo fertility preservation before receiving anti-tumor treatment and non-cancer patients who undergo assisted reproductive technology treatment/natural pregnancy.

This study will be conducted in the Clinical Center of Reproductive Medicine, First Affiliated Hospital of Nanjing Medical University. 2800 women diagnosed with malignant cancers who has desire to reproduce will be enrolled in this study.

Statistical analysis of the data will be performed.

DETAILED DESCRIPTION:
The number of new cancer cases among Chinese women in 2020 will be 2.09 million, showing a trend in younger age at the time of diagnosis. Incomplete statistics show that 25%~30% of young breast cancer patients in China Need for fertility preservation. In this study, we want to answer the question: Does fertility preservation affect the prognosis in female cancer patients.

This study will be conducted in the Clinical Center of Reproductive Medicine, First Affiliated Hospital of Nanjing Medical University. 2800 women diagnosed with malignant cancers who has desire to reproduce will be enrolled in this study.

If a female tumor patients (focusing on: breast cancer, hematological diseases/lymphoma, gynecological tumors (ovarian borderline tumors, etc.), nasopharyngeal cancer, colorectal cancer, etc.) have a desire to reproduce in the future, she would considered for enrollment. After being admitted into this study, according to the patients'own will, she will receive long term observation or fertility preservation followed by long term observation. Cumulative live birth rate, perinatal and perinatal complications, and offspring health of women who have or have not received fertility preservation before anti-tumor treatment and who have no tumor and who normally receive assisted reproductive technology treatment/natural pregnancy are all recorded, to assess the impact of the current new anti-tumor treatment on female fertility and offspring health.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor confirmed (main focus: breast cancer, hematological disease/lymphoma, gynecological tumor (ovarian cancer), boundary tumors, nasopharyngeal cancer, colorectal cancer, and other tumors that require anti-tumor treatment;
2. Having a desire for future fertility(including women who have already given birth);
3. Age: 20-40 years old (patients planning to freeze their eggs are ≤35 years old, and those planning to freeze their embryos are ≤40 years old);
4. Consent.

Exclusion Criteria:

1. Patients with congenital or acquired uterine abnormalities, severe intrauterine adhesions, and other diseases that have a clear impact on pregnancy;
2. Those with assisted reproductive technology and pregnancy contraindications;
3. Tumors that are not suitable for pregnancy after multidisciplinary discussions on tumor fertility;
4. Clinical diagnosis of POI (premature ovarian insufficiency).

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Female patients
Study Population: 2800 female cancer patients who have fertility desire
Sampling Method: Non-Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2032-10-01 (Estimated)

PRIMARY OUTCOMES:
5-year cumulative live birth rate | 5 years
  5-year cumulative live birth rate for female patients who reproduce

SECONDARY OUTCOMES:
Ovarian function(AMH levels) | 5 years
  AMH levels of all patients
Ovarian function(AFC counts) | 5 years
  AFC counts of of all patients
Newborn malformation rate | 5 years
  Newborn malformation rate for female patients who reproduced
Tumor recurrence rate | 5 years
  Tumor recurrence rate of all participants
Tumor survival rate | 5 years
  Tumor survival rate of all participants

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Center of Reproductive Medicine of First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol can be shared
Supporting Information: Study Protocol
Time Frame: 5 years